CLINICAL TRIAL: NCT03062228
Title: Korle Bu Teaching Hospital - Global Innovations for Reproductive Health & Life Healthy Birth Weight Study: A Cross-Section
Brief Title: KBTH-GIRHL Healthy Birth Weight Study: A Cross-Section
Acronym: KBTH-HBWS
Status: Completed | Type: Observational
Sponsor: IWK Health Centre (Other)
Collaborators: Korle Bu Teaching Hospital (Unknown); University of Michigan (Other); Innovative Canadians for Change (Other); Dalhousie University (Other); Global Innovations for Reproductive Health & Life (Unknown); University of Ghana Medical School (Other)
Responsible Party: Principal Investigator, Allan Kember, Medical Student, IWK Health Centre
Other Study IDs: KBTH-IRB/00020/2016
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Infant, Small for Gestational Age; Infant, Low Birth Weight; Pregnancy; Sleep; Infant, Very Low Birth Weight; Fetal Growth Retardation
Keywords: stillbirth; sleep; low birth weight; pregnancy; supine; small for gestational age
MeSH Terms: conditions — Fetal Growth Retardation; Stillbirth; Deception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Controls: Healthy, Ghanaian women who have recently delivered a live birth at the Korle Bu Teaching Hospital.
  No interventions will be administered.

SUMMARY:
This study was designed and conducted in an effort to establish a comparison group for the Ghana PrenaBelt Trial (NTC02379728). The Ghana PrenaBelt Trial examined the effect, on birth weight, of a belt-like device to help pregnant women to avoid sleeping on their back during sleep in the third trimester. This study will seek to establish the typical birth weight of babies born to a cohort of healthy pregnant Ghanian women who are similar in characteristics to the women in the Ghana PrenaBelt Trial but who have not been educated to avoid back sleep during pregnancy nor have received a device to prevent back sleep.

DETAILED DESCRIPTION:
Recently, three studies have suggested that maternal back sleep may be a risk factor for stillbirth (SB) and low birth weight (LBW). This is significant given that the majority of third-trimester pregnant women spend up to 25% of their sleep time on their back. The Ghana PrenaBelt Trial (GPT), completed by our team at the Korle Bu Teaching Hospital (KBTH) from September 2015 - May 2016, was the first interventional trial investigating this possible relationship between maternal back sleep and LBW. However, a limitation of the GPT was that due to its sham-control design, all participants in the trial (treatment group and sham-control group) were educated during the consent process about back-sleep in late pregnancy as a possible risk factor for SB and LBW. At interim analysis of the GPT (February 2016), no difference in birth weight was found between the two groups. Also around this time, the study team had anecdotal reports from sham-group participants who indicated that they trained themselves to sleep exclusively on their left side. Further, there is evidence in the literature that when instructed to sleep on their left, third-trimester pregnant women can increase the percentage of left-sided sleep to approximately 60% of the night on average and maintain this across multiple nights.

Given this, it was questioned if the back-sleep education during the consent process could be having an effect on the sleep behaviour of the GPT participants independently of their treatment allocation; therefore, the KBTH-GIRHL Healthy Birth Weight Study was designed in March 2016 to investigate this question further. The aim of this study is to establish a reference birth weight of babies born to a cohort of women comparable to the cohort in the GPT but who have not received back-sleep education, did not participate in the GPT, and whose babies were born in a similar time period and weighed on the same newborn scales - in essence, a control group for the GPT.

This cross-sectional study will be accomplished via recruiting a control group from a pool of women having recently delivered at KBTH, reviewing their hospital records, and having them complete a short survey about their demographics, obstetric history, and sleep behaviors.

The results of this study, together with the results of the GPT, will enable us to determine whether or not education about back-sleep in pregnancy affects pregnancy outcomes, specifically birth weight.

ELIGIBILITY:
Inclusion Criteria:

* Low-risk singleton pregnancy
* *Delivered a live birth >28 weeks gestation at KBTH within the past 48 hours.
* Residing in the Greater Accra Metropolitan Area or area served by the KBTH.
* Fluent in either English, Twi, or Ga
* **Has not received education/ information about back sleep position in pregnancy as a potential risk factor for stillbirth and low birth weight.

Exclusion Criteria:

* BMI ≥ 35 at booking (first antenatal appointment for current pregnancy)
* Pregnancy complicated by obstetric complications (hypertension [pre-eclampsia, gestational hypertension, chronic hypertension], diabetes [gestational or not], or intra-uterine growth restriction [<10th %ile for growth])
* Sleep complicated by medical conditions (known to get <4 hours of sleep per night due to insomnia, or musculoskeletal disorder that prevents sleeping on a certain side [e.g., arthritic shoulder])
* Multiple pregnancy
* Known fetal abnormality
* Maternal age >35

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants (subjects) will be healthy, Ghanaian women who have recently delivered a live birth at KBTH. The inclusion/exclusion criteria criteria will be similar to the Ghana PrenaBelt Trial with one difference (* below) and one additional inclusion criterion (** below).
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxfield Okere, B.Sc., Principal Investigator — Korle Bu Teaching Hospital
Locations (1):
- Korle Bu Teaching Hospital, Korle Bu, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owusu JT, Anderson FJ, Coleman J, Oppong S, Seffah JD, Aikins A, O'Brien LM. Association of maternal sleep practices with pre-eclampsia, low birth weight, and stillbirth among Ghanaian women. Int J Gynaecol Obstet. 2013 Jun;121(3):261-5. doi: 10.1016/j.ijgo.2013.01.013. Epub 2013 Mar 15. PMID 23507553
- [Background] Stacey T, Thompson JM, Mitchell EA, Ekeroma AJ, Zuccollo JM, McCowan LM. Association between maternal sleep practices and risk of late stillbirth: a case-control study. BMJ. 2011 Jun 14;342:d3403. doi: 10.1136/bmj.d3403. PMID 21673002
- [Background] Gordon A, Raynes-Greenow C, Bond D, Morris J, Rawlinson W, Jeffery H. Sleep position, fetal growth restriction, and late-pregnancy stillbirth: the Sydney stillbirth study. Obstet Gynecol. 2015 Feb;125(2):347-355. doi: 10.1097/AOG.0000000000000627. PMID 25568999
- [Background] Platts J, Mitchell EA, Stacey T, Martin BL, Roberts D, McCowan L, Heazell AE. The Midland and North of England Stillbirth Study (MiNESS). BMC Pregnancy Childbirth. 2014 May 21;14:171. doi: 10.1186/1471-2393-14-171. PMID 24885461
- [Background] Warland J, Mitchell EA. A triple risk model for unexplained late stillbirth. BMC Pregnancy Childbirth. 2014 Apr 14;14:142. doi: 10.1186/1471-2393-14-142. PMID 24731396
- [Background] O'Brien LM, Warland J. Typical sleep positions in pregnant women. Early Hum Dev. 2014 Jun;90(6):315-7. doi: 10.1016/j.earlhumdev.2014.03.001. Epub 2014 Mar 21. PMID 24661447
- [Background] Stone PR, Burgess W, McIntyre JP, Gunn AJ, Lear CA, Bennet L, Mitchell EA, Thompson JM; Maternal Sleep In Pregnancy Research Group, The University of Auckland. Effect of maternal position on fetal behavioural state and heart rate variability in healthy late gestation pregnancy. J Physiol. 2017 Feb 15;595(4):1213-1221. doi: 10.1113/JP273201. Epub 2016 Dec 11. PMID 27871127
- [Background] Warland J, Dorrian J. Accuracy of self-reported sleep position in late pregnancy. PLoS One. 2014 Dec 23;9(12):e115760. doi: 10.1371/journal.pone.0115760. eCollection 2014. PMID 25535960
- [Background] Gardosi J, Chang A, Kalyan B, Sahota D, Symonds EM. Customised antenatal growth charts. Lancet. 1992 Feb 1;339(8788):283-7. doi: 10.1016/0140-6736(92)91342-6. PMID 1346292
- [Background] Gardosi J, Mongelli M, Wilcox M, Chang A. An adjustable fetal weight standard. Ultrasound Obstet Gynecol. 1995 Sep;6(3):168-74. doi: 10.1046/j.1469-0705.1995.06030168.x. PMID 8521065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between April 28 2016 through February 22 2017, inclusive. Participants were recruited by the study recruiter from a sample of healthy, Ghanaian women presenting to the KBTH maternity wards and who delivered a live birth within the past 48 hours.
Pre-assignment Details: There were no significant events in the study after participant enrollment but prior to assignment to an arm or group. Two participants who were recruited were excluded from the study after it was discovered later that they did not fully meet the eligibility criteria (both had delivered stillborn infants).
Period: Overall Study
Arm/Group | Controls
Started | 162
Completed | 162
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Controls
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ghanaian | 162
Region of Enrollment [Count of Participants; unit: Participants]
  Ghana | 162
Gravidity [Count of Participants; unit: Participants]
  Gravida 1 | 33
  Gravida ≥2 | 129
Parity [Count of Participants; unit: Participants]
  Para 1 | 44
  Para ≥2 | 118
Education level [Count of Participants; unit: Participants]
  Tertiary | 21
  Vocational | 1
  Senior High | 52
  Junior High | 57
  Primary | 30
  Undisclosed | 1
Household Income [Mean (Standard Deviation); unit: Cedis per month] — Average currency exchange rate for recruitment period: 1 United States Dollar (USD) = 4.04 Cedis Population: Two participants did not wish to disclose this information.
  Cedis per month
    number analyzed (Participants) | 160
    (all) | 1144 (665)
BMI upon entering third trimester for current pregnancy [Mean (Standard Deviation); unit: kg/m^2] — This is the participants BMI in the period between 26 and 30 weeks' gestation for the current pregnancy.
  kg/m^2 | 27.7 (4.1)
Pre-pregnancy BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI at the beginning of the current pregnancy
  kg/m^2 | 25.8 (3.9)
Nightly sleep duration [Mean (Standard Deviation); unit: hours] — This is the participant's self-reported average nightly sleep duration in the past week.
  hours | 8.3 (1.5)
In the last week, sleep onset position [Count of Participants; unit: Participants]
  Left | 75
  Supine | 11
  Right | 76
  Prone | 0
In the last week, waking position [Count of Participants; unit: Participants]
  Left | 67
  Supine | 25
  Right | 70
  Prone | 0
When not pregnant, sleep onset position [Count of Participants; unit: Participants]
  Left | 1
  Supine | 87
  Right | 24
  Prone | 50
When not pregnant, waking position [Count of Participants; unit: Participants]
  Left | 0
  Supine | 97
  Right | 31
  Prone | 34
Part of bed sleeps on [Count of Participants; unit: Participants]
  Left | 50
  Right | 108
  Center | 1
  Other | 3
Pillow use [Count of Participants; unit: Participants]
  None | 16
  Under head | 146
  Between knees | 1
  Under tummy | 0
  Behind back | 0
  Pregnancy pillow | 0
  Under feet | 37
  Under legs | 0
Sleeps with bed partner [Count of Participants; unit: Participants] | 119
Uses insecticide treated bed net [Count of Participants; unit: Participants] | 50
Snores ≥3 nights per week [Count of Participants; unit: Participants] | 12
Past medical complications [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Birth Weight of Baby
Description: At delivery, birth weight will be measured and recorded in the participant's health record as a part of routine obstetric care at the Korle Bu Teaching Hospital.
Time Frame: Within 48 hours of delivery of baby (on average, 38 - 40 weeks gestation)
Population: Healthy, Ghanaian women who had recently (within 48 hours) delivered a live birth at the Korle Bu Teaching Hospital.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Controls
Number analyzed (Participants) | 162
grams | 3033 (514)

2. Primary Outcome: Customized Birth Weight Centile
Description: Individual customized birth weight centile calculated using the Gestation Network (Perinatal Institute; Birmingham, UK) Bulk Centile Calculator (BCC), which calculates customized birthweight centiles using the principles of the Gestation Related Optimal Weight (GROW) method.
  The main non-pathological factors affecting birth weight are gestational age, maternal height, maternal weight at booking, parity, and ethnic group. The sex of fetus/neonate, when known, should also be adjusted for. These six variables need to be adjusted for to calculate the true growth potential, which can be represented as individually customized fetal growth curves and birth weight percentiles using the principles of the GROW. This method for calculating growth potential has been validated in a number of international studies.
Time Frame: Within 48 hours of delivery of baby (on average, 38 - 40 weeks gestation)
Population: Healthy, Ghanaian women who had recently (within 48 hours) delivered a live birth at the Korle Bu Teaching Hospital.
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Controls
Number analyzed (Participants) | 162
percentile | 46.0 (30.5)

3. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age at delivery (weeks) will be recorded in the participant's health record as a part of routine obstetric care at the Korle Bu Teaching Hospital.
Time Frame: Within 48 hours of delivery of baby (on average, 38 - 40 weeks gestation)
Population: Healthy, Ghanaian women who had recently (within 48 hours) delivered a live birth at the Korle Bu Teaching Hospital.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Controls
Number analyzed (Participants) | 162
Weeks | 38.3 (2.5)

4. Secondary Outcome: Small for Gestational Age
Description: Small for Gestational Age is defined as a birthweight centile ≤10th centile per the Gestation-Related Optimal Weight (GROW) standard.
Time Frame: Within 48 hours of delivery of baby (on average, 38 - 40 weeks gestation)
Population: Healthy, Ghanaian women who had recently (within 48 hours) delivered a live birth at the Korle Bu Teaching Hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Controls
Number analyzed (Participants) | 162
Participants | 25

5. Secondary Outcome: Low Birth Weight
Description: Low birth weight is defined has birth weight ≤ 2500 grams.
Time Frame: Within 48 hours of delivery of baby (on average, 38 - 40 weeks gestation)
Population: Healthy, Ghanaian women who had recently (within 48 hours) delivered a live birth at the Korle Bu Teaching Hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Controls
Number analyzed (Participants) | 162
Participants | 21

6. Secondary Outcome: Sex of Newborn
Description: Sex of participant's newborn.
Time Frame: Within 48 hours of delivery of baby (on average, 38 - 40 weeks gestation)
Population: Healthy, Ghanaian women who had recently (within 48 hours) delivered a live birth at the Korle Bu Teaching Hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Controls
Number analyzed (Participants) | 162
Participants
  Male | 82
  Female | 80

7. Secondary Outcome: Preterm Delivery
Description: Preterm delivery is defined as gestational age at birth <37 weeks.
Time Frame: Within 48 hours of delivery of baby (on average, 38 - 40 weeks gestation)
Population: Healthy, Ghanaian women who had recently (within 48 hours) delivered a live birth at the Korle Bu Teaching Hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Controls
Number analyzed (Participants) | 162
Participants | 42

8. Secondary Outcome: Mode of Delivery
Description: Mode of delivery (spontaneous vaginal, Cesarean section, instrumented) will be recorded in the participant's health record as a part of routine obstetric care at the Korle Bu Teaching Hospital.
Time Frame: Within 48 hours of delivery of baby (on average, 38 - 40 weeks gestation)
Population: Healthy, Ghanaian women who had recently (within 48 hours) delivered a live birth at the Korle Bu Teaching Hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Controls
Number analyzed (Participants) | 162
Participants
  Spontaneous vaginal | 122
  Caesarean section | 40
  Instrumented | 0

ADVERSE EVENTS:
Time Frame: From delivery of infant (spontaneous vaginal delivery, instrumented vaginal delivery, cesarean section delivery) through discharge of the participant from hospital, which was 24 hours for a spontaneous vaginal delivery and 48 hours for an instrumented vaginal delivery or cesarean section delivery.
Arm/Group | Controls
All-Cause Mortality (participants affected / at risk) | 0/162
Serious Adverse Events (participants affected / at risk) | 0/162
Other Adverse Events (participants affected / at risk) | 0/162

LIMITATIONS AND CAVEATS:
Reliance on participant's self reports for some baseline characteristics data (e.g., pre-pregnancy BMI, sleep positions).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03062228/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03062228/SAP_001.pdf